CLINICAL TRIAL: NCT06880991
Title: Development of Patient-Reported Outcome Measures Assessing Tumor Visibility and Appearance Concerns in Neurofibromatosis Type 1: A Qualitative Study
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002268; 002268-C
Record Dates: First submitted 2025-03-15; First posted 2025-03-18 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09-25

CONDITIONS: Neurofibromatosis Type 1; Neurofibroma
Keywords: Qualitative; Focus Groups; Instrument Development
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1, Participants with pNF: Individuals age 8+ years with plexiform neurofibroma (pNF) tumor
  Interventions: Other: Arm 1
- Cohort 2, Caregiver of children with pNF: Caregivers of children (ages 5-17 years) with a plexiform neurofibroma (pNF) tumor
  Interventions: Other: Arm 1
- Cohort 3, Participants with cNF: Individuals age 12+ years with cutaneous neurofibroma (cNF) tumors
  Interventions: Other: Arm 1
- Cohort 4, Caregiver of children with cNF: Caregivers of children (ages 12-17 years) with cutaneous neurofibroma (cNF) tumors
  Interventions: Other: Arm 1

INTERVENTIONS:
Other: Arm 1 — Participant completion of questionnaires and participation in focus group(s) and/or interview sessions.

SUMMARY:
Background:

Neurofibromatosis 1 (NF1) is a disease that causes tumors to grow along the nerves. These include plexiform neurofibromas (pNF) and cutaneous neurofibromas (cNF). Both pNF and cNF can be visible to other people. These tumors can affect a person s appearance and quality of life. Researchers want to be able to assess changes in appearance before and after treatment for NF1 tumors.

Objective:

To see if two questionnaires can help assess people s ratings about the appearance of their pNF and cNF tumors.

Eligibility:

People aged 8 years and older with pNF and people 12 years and older either with cNF or both pNF and cNF. Adult caregivers of children with pNF and cNF are also needed.

Design:

Participants will complete questionnaires on paper or by phone, computer, or tablet. They will answer questions about how they look, how they feel, and how they feel about the way they look.

Participants will meet in at least 1 remote focus group or individual interview. The meeting will last about 1 hour. Each group will include 3 to 5 people, organized by age: 8 to 11 years, 12 to 17 years, 18 to 29 years, and over 30 years. Adult caregivers will meet in a group with other caregivers.

They will discuss their NF1 symptoms; how their tumors look; how they feel about the way their tumors look; and their daily activities. They will give their opinions about 2 questionnaires about appearance.

The group and individual meetings will be audio-recorded and transcribed. Information that can reveal individual identities will be removed.

DETAILED DESCRIPTION:
Background:

* Individuals with neurofibromatosis type 1 (NF1) may develop plexiform neurofibroma (pNF) and cutaneous neurofibroma (cNF) tumors, both of which can impact one s physical appearance and quality of life.
* To date, there are no validated patient-reported outcome (PRO) measures to assess tumor visibility or appearance-related concerns for individuals with these tumors.
* The Response Evaluation in Neurofibromatosis and Schwannomatosis (REiNS) PRO working group, which includes professionals from multiple disciplines and patient representatives, has reviewed disfigurement and appearance concerns measures for potential use in pNF and cNF clinical research trials.
* The group modified existing items to create the Tumor Visibility Rating Scale (TVRS) for pNF (TVRS-pNF) and TVRS for cNF tumors (TVRS-cNF).
* Among measures of appearance concerns reviewed by the REiNS PRO group, the FACEQ was the top candidate for use in NF1 clinical trials but will need to be qualitatively analyzed to confirm its appropriateness.

Primary Objective:

-To evaluate newly developed measures of tumor visibility (TVRS-pNF and TVRS-cNF) and to select the most appropriate items to assess these constructs in NF1 based on qualitative feedback from children and adults with NF1 and caregivers of children with NF1 to use as endpoints in clinical trials

Eligibility:

* Age 8 plus years for pNF tumors and 12 plus years for cNF tumors
* Self-reported diagnosis of NF1 with a pNF and/or cNF tumor(s) or caregiver of a child with NF1 with visible pNF and/or cNF tumor(s)
* Comfortable discussing their medical condition in English
* Access to a device with internet

Design:

* This is a qualitative study that seeks to enroll children and adults with pNF and/or cNF tumors and caregivers of a child with these tumors to take part in focus groups and interviews about the domains and measures of interest. These results will inform modifications to the measures.
* A sample size of 90 participants is expected to be sufficient to meet our objectives. To account for inevaluable participants, the accrual ceiling is 110.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must self-report a diagnosis of NF1 OR be the caregiver of a child with NF1 (5-17 years old with plexiform neurofibroma [pNF] or 12-17 years old with cutaneous neurofibroma [cNF])

The following for the participant or the caregiver of a child, as appropriate:

* Participants with NF1 must self-report a pNF and/or cNF tumor(s) that is visible to that individual OR others
* Caregivers of a child with NF1 must report a pNF and/or cNF tumor(s) that the child has that is visible to the child OR others
* Age requirements:

  * >= 8 years old (participants with pNF)
  * >= 12 years old (participants with cNF)
  * >= 12 years old (participants with pNF and cNF)
  * >= 18 years (caregivers)
* Access to device with internet
* Ability to understand English and comfort discussing their medical condition in English
* The ability of adult participant or caregiver of minor participants to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

* Physical or cognitive limitations that would prevent them from being able to participate in a focus group or interview, or unwillingness to do so
* Since we will aim to have no less than 25 percent of participants from underrepresented* groups, individuals from represented groups may not be able to participate after we have reached the maximum target for represented groups. Consistent with best practices for scale development and validation, this will help ensure that the measures are appropriate for people from a variety of backgrounds.

  * Underrepresented groups are defined as people who identify as African American or Black, American Indian, Alaska Native, Hispanic/Latine, Native Hawaiian, and other Pacific Islander.
* If saturation has been met within a particular age group, potential participants from that completed age group will no longer be eligible.

Ages: 5 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: individuals with neurofibromatosis type 1 (NF1) or be the caregiver of a child with NF1 (5-17 years old with plexiform neurofibroma [pNF] or 12-17 years old with cutaneous neurofibroma [cNF]).
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate new tumor visibility (DRS-pNF, DRS-cNF self-report/parent-report); to select the most appropriate items to assess these constructs in NF1 based on qualitative feedback from children and adults with NF1 and visible pNF or cNF | throughout the study
  The primary endpoints will be the modified measures of tumor visibility resulting from the qualitative data obtained from the focus groups and interviews.

SECONDARY OUTCOMES:
Evaluate an existing measure of appearance concerns based on qualitative feedback from children & adults with NF1 and visible pNF and/or cNF tumors and caregivers of children with NF1 to determine its appropriateness for NF1 clinical tri... | throughout the study
  The secondary endpoint will be either the FACE-Q or a newly developed measure of appearance concerns, depending on the results of the qualitative focus groups and interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Staci M Peron, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared after completion of the primary endpoint per the data management sharing plan.
Access Criteria: Data may be requested by contacting the Principal Investigator.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002268-C.html